CLINICAL TRIAL: NCT06953284
Title: Efficacy of Kinesiotaping Versus Functional Electrical Stimulation on Equinus Deformity in Children With Diplegic Cerebral Palsy
Brief Title: Kinesiotaping Versus Functional Electrical Stimulation on Equinus Deformity
Acronym: KINESOTAPING
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Sara Yousef Abdel Elglil Yousef Elsebahy, lecturer of physical therapy for pediatrics, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-496
Record Dates: First submitted 2025-04-12; First posted 2025-05-01 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: EQUINUS DEFORMITY
Keywords: KINESOTAPING; FUNCTIONAL ELECTRICAL STIMULATION; EQUINUS DEFORMITY; DIAPLEGIC CEREBRAL PALSY
MeSH Terms: conditions — Equinus Deformity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): children will receive kinesiotap technique in addition to the designed physiotherapy program for 3 months 3 session per week
  Interventions: Other: KINESOTAPING
- group 2 (Experimental): children will receive FUNCTIONAL ELECTRICAL STIMULATION in addition to the designed physiotherapy program for 3 months 3session per week
  Interventions: Other: Functional Electrical Stimulation

INTERVENTIONS:
Other: KINESOTAPING — Kinesio Taping (KT) is commonly used in sport injuries, in neurology and oncology patients following the surgical protocols, and for paediatric rehabilitation to reduce pain, facilitate or inhibit muscle activity, prevent injuries, reposition joints, aid the lymphatic system, support postural alignment, and improve proprioception.7-9 Although its mechanism of action has not been fully understood, it is believed that activation of the cutaneous receptors could influence neuromuscular functions.10 The cutaneous sensory system provides preliminary information about limb positions and muscle forces to the central nervous system for monitoring and controlling limb movements, planning actions, and providing fluent movement.11 Common causes of unilateral spastic CP are middle cerebral artery infarct, hemi-brain atrophy, periventricular lesions, and brain malformations that disturb the integrity of the motor areas. Middle cerebral artery infarctions can particularly impair the somatosensory sy
  Arms: group 1
Other: Functional Electrical Stimulation — This systematic review is the first to examine the effect of FES on activity in children with CP using only randomized trials.However, evidence was limited with only 5 trials being included. This limited evidence suggests that FES is effective, that is, it is better than no FES intervention, but that it is no more effective than activity training, that is, practicing the activity without FES will be just as effective. Furthermore, no evidence was found on whether any benefits are maintained beyond the intervention period because even though a follow-up measurement was reported for 2 studies, the authors failed to provide data. Even though the review was restricted to the highest standard of evidence, randomized trials, firm conclusions cannot be made. This is primarily because of the absence of group data (means and SD) in the papers, preventing a meta-analysis. This poor reporting is disappointing given that 3 of the 5 trials were published within the last 5 years. Therefore, we may b
  Arms: group 2

SUMMARY:
Effect of FES Versus No FES intervention. A statistically significant between-group difference in activity in favor of FES was reported for all 3 studies, immediately after the intervention period. This difference represented a 30% to 32% greater increase in activity compared with no FES intervention. A follow-up measurement was reported for 1 study, but no data were reported.

Effect of FES Versus Activity Training. Both studies reported a statistically nonsignificant between-group difference in activity compared with activity training, immediately after the intervention period. One study included a follow-up measurement, but no data were reported

DETAILED DESCRIPTION:
This study will be conducted at the Outpatient clinics, Faculty of Physical

Therapy Kafrelsheikh University to prove the effect of core stability exercises on standing , balance and gait in diplegic CP children.

the children will be randomly allocated by simple random method via choosing one of two wrapped cards representing the two treatment groups, which are: Group (A): will receive core stability exercises in addition to the designed physiotherapy program.

Group (B): will receive the designed physiotherapy program only . Inclusion criteria

Children will be included in the study if they fulfil the following criteria:

1. A medical diagnosis of diplegic CP made by paediatricians or pediatric neurologists.
2. Children with spasticity grades ranged from 1 to 1+ according to MAS.
3. Their age range from 4 to 10 years.

1. Children were level I or II on the Gross Motor Function Classifcation System (GMFCS) 5.No orthopedic surgeries.

Exclusion criteria

Children will be excluded from the study if:

1. They had a permanent deformity (bony or soft tissue contractures).
2. Children having visual or auditory defects.
3. Children who had Botox application to the lower extremity in the past 6 months or had undergone a previous surgical intervention to ankle and knee.
4. A history of epileptic seizure and any diagnosed cardiac or orthopaedic disability that may prevent the use of assessment methods.
5. Children who are absent in two successive sessions.

ELIGIBILITY:
Inclusion Criteria:

* 1. A medical diagnosis of diplegic CP made by paediatricians or pediatric neurologists.

  2. Children with spasticity grades ranged from 1 to 1+ according to MAS. 3. Their age range from 4 to 10 years.
  1. Children were level I or II on the Gross Motor Function Classifcation System (GMFCS) 5.No orthopedic surgeries

     Exclusion Criteria:

  <!-- -->

  1. They had a permanent deformity (bony or soft tissue contractures).
  2. Children having visual or auditory defects.
  3. Children who had Botox application to the lower extremity in the past 6 months or had undergone a previous surgical intervention to ankle and knee.
  4. A history of epileptic seizure and any diagnosed cardiac or orthopaedic disability that may prevent the use of assessment methods.
  5. Children who are absent in two successive sessions.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
1. balance | 3 months
  pediatric balance scale is clinical assessment tool designed to evaluate functional balance in children, particularly those with motor impairments such as cerebral palsy or developmental delays. It is a modified version of the Berg Balance Scale, adapted to suit the functional capabilities and developmental stages of children aged approximately 2 to 15 years.
2. Evaluation of gait | 3 months
  Kinovea is a free, open-source video analysis software widely used in clinical and research settings for the assessment of human movement, including gait analysis. It allows for detailed observation and measurement of kinematic parameters, such as joint angles, stride length, step time, and gait symmetry, through frame-by-frame video playback and annotation tools. To assess gait, videos of a subject walking are captured using a standard camera and then imported into Kinovea. The software enables users to place markers on key anatomical landmarks, which can then be tracked throughout the gait cycle
3. Evaluation of standing | 3 months
  The Gross Motor Function Classification System (GMFCS) is a standardized tool used to evaluate and classify the gross motor function of children with cerebral palsy, focusing on self-initiated movements, particularly in sitting and walking. It consists of five levels (I to V), with Level I indicating the most independent motor function and Level V the most severe limitations. In the context of evaluating standing progress, the GMFCS provides a reliable framework to monitor changes in a child's ability to maintain or achieve standing posture over time. For example, a transition from requiring support to stand (Level IV or III) to standing independently or with minimal assistance (Level II or I) reflects significant motor improvement. The classification system is age-specific and considers developmental milestones, making it especially useful for tracking functional gains during rehabilitation or intervention programs. Its ease of use, validity, and consistency make GMFCS an essential t

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided